CLINICAL TRIAL: NCT04683510
Title: Increasing Recruitment of Underrepresented Cancer Survivors With Awareness Enhancing Interventions
Brief Title: Awareness Enhancing Interventions
Acronym: AWEI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, MICHELLE Y MARTIN, Director: Center for Innovation in Health Equity Research, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 300002068-B; R01CA242737-01A1 (NIH)
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Research Awareness
Keywords: Cancer Survivors; African American; Awareness

STUDY DESIGN:
Intervention Model Description: AMPLIFI recruitment process, 1600 AA cancer survivors will be randomized to one of 8 conditions that vary by type of strategy, type of information, and type of perspective (survivor or researcher "voice") and 400 randomized to the basic recruitment strategy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): This group will receive no intervention before receiving the AMPLIFI Recruitment Call
- Navigation (Other): After receiving recruitment letter from AMPLIFI, participant randomized to this arm will receive a phone call from a Research Specialist who will discuss the importance of research participation for cancer survivors to increase research awareness and aid in recruitment. The information will focus on the importance of research and will be delivered from the perspective of either a researcher or a cancer survivor.
  Interventions: Other: Navigation - Study Specific - Researcher Voice; Other: Navigation - Study Specific - Cancer Survivor Voice; Other: Navigation - Research General - Researcher Voice; Other: Navigation - Research General - Cancer Survivor Voice
- Brochure (Other): After receiving recruitment letter from AMPLIFI, participant randomized to this arm will receive a brochure which will focus on the importance of research participation for cancer survivors in order to increase research awareness and aid in recruitment.
  Interventions: Other: Brochure - Study Specific - Researcher Voice; Other: Brochure - Study Specific - Cancer Survivor Voice; Other: Brochure - Research General - Researcher Voice; Other: Brochure - Research General - Cancer Survivor Voice

INTERVENTIONS:
Other: Navigation - Study Specific - Researcher Voice — The intervention is delivered over the telephone
  Arms: Navigation
Other: Navigation - Study Specific - Cancer Survivor Voice — The intervention is delivered over the telephone
  Arms: Navigation
Other: Navigation - Research General - Researcher Voice — The intervention is delivered over the telephone
  Arms: Navigation
Other: Navigation - Research General - Cancer Survivor Voice — The intervention is delivered over the telephone
  Arms: Navigation
Other: Brochure - Study Specific - Researcher Voice — The invention is mailed to the participant in a brochure.
  Arms: Brochure
Other: Brochure - Study Specific - Cancer Survivor Voice — The invention is mailed to the participant in a brochure.
  Arms: Brochure
Other: Brochure - Research General - Researcher Voice — The invention is mailed to the participant in a brochure.
  Arms: Brochure
Other: Brochure - Research General - Cancer Survivor Voice — The invention is mailed to the participant in a brochure.
  Arms: Brochure

SUMMARY:
The purpose of this study is to determine if increasing awareness and, thus, enhancing positive attitudes about research, prior to recruitment attempts, will increase participation in cancer clinical research among African American (AA) cancer survivors so that recruitment efforts can focus on the most optimal and cost- effective approaches

DETAILED DESCRIPTION:
In this project, 2000 AA potential AMPLIFI project participants will be randomized to the awareness-enhancing intervention (AWEI) or to the comparison condition in which they do not receive AWEI intervention but only the Adapting Multiple Behavior Interventions that Effectively Improve Cancer Survivor Health (AMPLIFI) basic recruitment strategy (No AWEI). Randomization for the AWEI Randomized Controlled Trial (RCT) will occur soon after the AMPLIFI recruitment letter is sent, and AWEI interventions will be delivered over a two-week period between the AMPLIFI recruitment invitation letter and the AMPLIFI recruitment call. Survivors randomized to AWEI intervention will be exposed to 8 different combinations of the AWEI components according to different types of strategies and type of information reflecting the survivor voice or not. Subsequent to the AMPLIFI recruitment call, a 20% random sample of cancer survivors will be surveyed over the phone to assess intervention fidelity.

ELIGIBILITY:
Inclusion Criteria:

* African American/Black
* adults (age ≥50 years old)
* diagnosed with obesity/physical activity associated cancers that have a 70% or greater 5-year relative cancer-free survival rate multiple myeloma, localized kidney cancer and loco- regional cancers of the colorectum, female breast, prostate, endometrium, and ovary).
* 1-5 years post diagnosis
* reside in an area with wireless coverage
* In the AMPLIFI recruitment pool

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4451 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Y Marttin, PhD, Principal Investigator — University of Tennessee; Maria Pisu, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Tennessee Health Science Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
We will share data which will include the AMPLIFI final disposition code (recruited versus not recruited), the impact of the AWEI interventions versus the standard recruitment approach.
Supporting Information: Study Protocol, SAP
Time Frame: All data will be shared once all primary outcomes papers have been published (consonant with the NIH definition of "timely fashion") but no later than within one year of the completion of the funded study.
Access Criteria: The access to the data will be granted to investigators working in an organization with a Federal Wide Assurance (FWA). Before access is granted, individuals must provide a copy of their Institutional Review Board (IRB) approval to use the data to answer their specific study questions. Individuals in receipt of data must produce proof of human subjects and HIPAA training. All datasets will conform to the "Standards for Privacy of Individually Identifiable Health Information" rule of HIPAA. In order to maintain HIPAA compliance, we will provide a limited-use dataset (i.e., stripped of identifying information). Requesting users will be required to sign a data-use sharing agreement. Although not immediately precluded, data deemed to be "sensitive" will be added to limited use datasets only after careful consideration. Resulting publications must credit the funding for this grant.

REFERENCES:
- [Background] Bester N, Di Vito-Smith M, McGarry T, Riffkin M, Kaehler S, Pilot R, Bwire R. The Effectiveness of an Educational Brochure as a Risk Minimization Activity to Communicate Important Rare Adverse Events to Health-Care Professionals. Adv Ther. 2016 Feb;33(2):167-77. doi: 10.1007/s12325-016-0284-y. Epub 2016 Jan 23. PMID 26801772
- [Background] Beskow LM, Sandler RS, Millikan RC, Weinberger M. Patient perspectives on research recruitment through cancer registries. Cancer Causes Control. 2005 Dec;16(10):1171-5. doi: 10.1007/s10552-005-0407-2. PMID 16215867
- [Background] Wenzel JA, Mbah O, Xu J, Moscou-Jackson G, Saleem H, Sakyi K, Ford JG. A Model of Cancer Clinical Trial Decision-making Informed by African-American Cancer Patients. J Racial Ethn Health Disparities. 2015 Jun;2(2):192-9. doi: 10.1007/s40615-014-0063-x. PMID 25960945
- [Background] Doak LG, Doak CC, Meade CD. Strategies to improve cancer education materials. Oncol Nurs Forum. 1996 Sep;23(8):1305-12. PMID 8883075
- [Background] Ford JG, Howerton MW, Bolen S, Gary TL, Lai GY, Tilburt J, Gibbons MC, Baffi C, Wilson RF, Feuerstein CJ, Tanpitukpongse P, Powe NR, Bass EB. Knowledge and access to information on recruitment of underrepresented populations to cancer clinical trials. Evid Rep Technol Assess (Summ). 2005 Jun;(122):1-11. doi: 10.1037/e439572005-001. No abstract available. PMID 15989377
- [Background] Hughes TB, Varma VR, Pettigrew C, Albert MS. African Americans and Clinical Research: Evidence Concerning Barriers and Facilitators to Participation and Recruitment Recommendations. Gerontologist. 2017 Apr 1;57(2):348-358. doi: 10.1093/geront/gnv118. PMID 26553736
- [Background] Kamen CS, Quinn GP, Asare M, Heckler CE, Guido JJ, Giguere JK, Gilliland K, Liu JJ, Geer J, Delacroix SE, Morrow GR, Jacobsen PB. Multimedia psychoeducation for patients with cancer who are eligible for clinical trials: A randomized clinical trial. Cancer. 2018 Dec 1;124(23):4504-4511. doi: 10.1002/cncr.31771. Epub 2018 Oct 6. PMID 30291797
- [Background] Fouad MN, Acemgil A, Bae S, Forero A, Lisovicz N, Martin MY, Oates GR, Partridge EE, Vickers SM. Patient Navigation As a Model to Increase Participation of African Americans in Cancer Clinical Trials. J Oncol Pract. 2016 Jun;12(6):556-63. doi: 10.1200/JOP.2015.008946. Epub 2016 May 17. PMID 27189356
- [Background] Ward EM, Sherman RL, Henley SJ, Jemal A, Siegel DA, Feuer EJ, Firth AU, Kohler BA, Scott S, Ma J, Anderson RN, Benard V, Cronin KA. Annual Report to the Nation on the Status of Cancer, Featuring Cancer in Men and Women Age 20-49 Years. J Natl Cancer Inst. 2019 Dec 1;111(12):1279-1297. doi: 10.1093/jnci/djz106. PMID 31145458
- [Background] Wissing MD, Kluetz PG, Ning YM, Bull J, Merenda C, Murgo AJ, Pazdur R. Under-representation of racial minorities in prostate cancer studies submitted to the US Food and Drug Administration to support potential marketing approval, 1993-2013. Cancer. 2014 Oct 1;120(19):3025-32. doi: 10.1002/cncr.28809. Epub 2014 Jun 25. PMID 24965506
- [Background] Shenoy D, Packianathan S, Chen AM, Vijayakumar S. Do African-American men need separate prostate cancer screening guidelines? BMC Urol. 2016 May 10;16(1):19. doi: 10.1186/s12894-016-0137-7. PMID 27165293
- [Background] Ewing AT, Kalu N, Cain G, Erby LH, Ricks-Santi LJ, Tetteyfio-Kidd Telemaque E, Scott DM. Factors associated with willingness to provide biospecimens for genetics research among African American cancer survivors. J Community Genet. 2019 Oct;10(4):471-480. doi: 10.1007/s12687-019-00411-0. Epub 2019 Mar 14. PMID 30877487
- [Background] Rivers D, August EM, Sehovic I, Lee Green B, Quinn GP. A systematic review of the factors influencing African Americans' participation in cancer clinical trials. Contemp Clin Trials. 2013 Jul;35(2):13-32. doi: 10.1016/j.cct.2013.03.007. Epub 2013 Apr 1. PMID 23557729
- [Background] Rick J, Graffy J, Knapp P, Small N, Collier DJ, Eldridge S, Kennedy A, Salisbury C, Treweek S, Torgerson D, Wallace P, Madurasinghe V, Hughes-Morley A, Bower P. Systematic techniques for assisting recruitment to trials (START): study protocol for embedded, randomized controlled trials. Trials. 2014 Oct 25;15:407. doi: 10.1186/1745-6215-15-407. PMID 25344684
- [Background] Treweek S, Lockhart P, Pitkethly M, Cook JA, Kjeldstrom M, Johansen M, Taskila TK, Sullivan FM, Wilson S, Jackson C, Jones R, Mitchell ED. Methods to improve recruitment to randomised controlled trials: Cochrane systematic review and meta-analysis. BMJ Open. 2013 Feb 7;3(2):e002360. doi: 10.1136/bmjopen-2012-002360. Print 2013. PMID 23396504
- [Background] Madurasinghe VW; Sandra Eldridge on behalf of MRC START Group and Gordon Forbes on behalf of the START Expert Consensus Group. Guidelines for reporting embedded recruitment trials. Trials. 2016 Jan 14;17:27. doi: 10.1186/s13063-015-1126-y. PMID 26767365
- [Background] Pisu M, Demark-Wahnefried W, Kenzik KM, Oster RA, Lin CP, Manne S, Alvarez R, Martin MY. A dance intervention for cancer survivors and their partners (RHYTHM). J Cancer Surviv. 2017 Jun;11(3):350-359. doi: 10.1007/s11764-016-0593-9. Epub 2017 Jan 9. PMID 28070770
- [Background] Martin MY, Pollack LA, Evans MB, Smith JL, Kratt P, Prayor-Patterson H, Watson CD, Dignan M, Cheney LC, Pisu M, Liwo A, Hullett S. Tailoring cancer education and support programs for low-income, primarily African American cancer survivors. Oncol Nurs Forum. 2011 Jan;38(1):E55-9. doi: 10.1188/11.ONF.E55-E59. PMID 21186152
- [Background] Pisu M, Martin MY, Shewchuk R, Meneses K. Dealing with the financial burden of cancer: perspectives of older breast cancer survivors. Support Care Cancer. 2014 Nov;22(11):3045-52. doi: 10.1007/s00520-014-2298-9. Epub 2014 Jun 10. PMID 24912858
- [Background] Pisu M, Azuero A, Halilova KI, Williams CP, Kenzik KM, Kvale EA, Williams GR, Meneses K, Sullivan M, Yagnik SK, Goertz HP, Rocque GB. Most impactful factors on the health-related quality of life of a geriatric population with cancer. Cancer. 2018 Feb 1;124(3):596-605. doi: 10.1002/cncr.31048. Epub 2017 Dec 18. PMID 29250775
- [Background] Pisu M, Schoenberger YM, Herbey I, Brown-Galvan A, Liang MI, Riggs K, Meneses K. Perspectives on Conversations About Costs of Cancer Care of Breast Cancer Survivors and Cancer Center Staff: A Qualitative Study. Ann Intern Med. 2019 May 7;170(9_Suppl):S54-S61. doi: 10.7326/M18-2117. PMID 31060056
- [Background] Martin MY, Evans MB, Kratt P, Pollack LA, Smith JL, Oster R, Dignan M, Prayor-Patterson H, Watson C, Houston P, Andrews S, Liwo A, Tseng TS, Hullett S, Oliver J, Pisu M. Meeting the information needs of lower income cancer survivors: results of a randomized control trial evaluating the american cancer society's "I can cope". J Health Commun. 2014 Apr;19(4):441-59. doi: 10.1080/10810730.2013.821557. Epub 2014 Jan 16. PMID 24433231
- [Background] Fouad M, Wynn T, Martin M, Partridge E. Patient navigation pilot project: results from the Community Health Advisors in Action Program (CHAAP). Ethn Dis. 2010 Spring;20(2):155-61. PMID 20503896
- [Background] Dignan M, Evans M, Kratt P, Pollack LA, Pisu M, Smith JL, Prayor-Patterson H, Houston P, Watson C, Hullett S, Martin MY. Recruitment of low income, predominantly minority cancer survivors to a randomized trial of the I Can Cope cancer education program. J Health Care Poor Underserved. 2011 Aug;22(3):912-24. doi: 10.1353/hpu.2011.0069. PMID 21841287
- [Background] Schoenberger YM, Benz R, McNees P, Meneses K. Patient-centered outcome evaluation of the Rural Breast Cancer Survivors Intervention. Support Care Cancer. 2016 Apr;24(4):1841-8. doi: 10.1007/s00520-015-2974-4. Epub 2015 Oct 9. PMID 26452487
- [Background] Demark-Wahnefried W, Case LD, Blackwell K, Marcom PK, Kraus W, Aziz N, Snyder DC, Giguere JK, Shaw E. Results of a diet/exercise feasibility trial to prevent adverse body composition change in breast cancer patients on adjuvant chemotherapy. Clin Breast Cancer. 2008 Feb;8(1):70-9. doi: 10.3816/CBC.2008.n.005. PMID 18501061
- [Background] Demark-Wahnefried W, Clipp EC, Lipkus IM, Lobach D, Snyder DC, Sloane R, Peterson B, Macri JM, Rock CL, McBride CM, Kraus WE. Main outcomes of the FRESH START trial: a sequentially tailored, diet and exercise mailed print intervention among breast and prostate cancer survivors. J Clin Oncol. 2007 Jul 1;25(19):2709-18. doi: 10.1200/JCO.2007.10.7094. PMID 17602076
- [Background] Demark-Wahnefried W, Clipp EC, Morey MC, Pieper CF, Sloane R, Snyder DC, Cohen HJ. Lifestyle intervention development study to improve physical function in older adults with cancer: outcomes from Project LEAD. J Clin Oncol. 2006 Jul 20;24(21):3465-73. doi: 10.1200/JCO.2006.05.7224. PMID 16849763
- [Background] Demark-Wahnefried W, Jones LW, Snyder DC, Sloane RJ, Kimmick GG, Hughes DC, Badr HJ, Miller PE, Burke LE, Lipkus IM. Daughters and Mothers Against Breast Cancer (DAMES): main outcomes of a randomized controlled trial of weight loss in overweight mothers with breast cancer and their overweight daughters. Cancer. 2014 Aug 15;120(16):2522-34. doi: 10.1002/cncr.28761. Epub 2014 May 7. PMID 24804802
- [Background] Adams RN, Mosher CE, Blair CK, Snyder DC, Sloane R, Demark-Wahnefried W. Cancer survivors' uptake and adherence in diet and exercise intervention trials: an integrative data analysis. Cancer. 2015 Jan 1;121(1):77-83. doi: 10.1002/cncr.28978. Epub 2014 Aug 25. PMID 25155573
- [Background] Durant RW, Wenzel JA, Scarinci IC, Paterniti DA, Fouad MN, Hurd TC, Martin MY. Perspectives on barriers and facilitators to minority recruitment for clinical trials among cancer center leaders, investigators, research staff, and referring clinicians: enhancing minority participation in clinical trials (EMPaCT). Cancer. 2014 Apr 1;120 Suppl 7(0 7):1097-105. doi: 10.1002/cncr.28574. PMID 24643647
- [Background] Demark-Wahnefried W, Bowen DJ, Jabson JM, Paskett ED. Scientific bias arising from sampling, selective recruitment, and attrition: the case for improved reporting. Cancer Epidemiol Biomarkers Prev. 2011 Mar;20(3):415-8. doi: 10.1158/1055-9965.EPI-10-1169. PMID 21382981
- [Background] Snyder DC, Morey MC, Sloane R, Stull V, Cohen HJ, Peterson B, Pieper C, Hartman TJ, Miller PE, Mitchell DC, Demark-Wahnefried W. Reach out to ENhancE Wellness in Older Cancer Survivors (RENEW): design, methods and recruitment challenges of a home-based exercise and diet intervention to improve physical function among long-term survivors of breast, prostate, and colorectal cancer. Psychooncology. 2009 Apr;18(4):429-39. doi: 10.1002/pon.1491. PMID 19117329
- [Background] Fowke JH, Schlundt D, Signorello LB, Ukoli FA, Blot WJ. Prostate cancer screening between low-income African-American and Caucasian men. Urol Oncol. 2005 Sep-Oct;23(5):333-40. doi: 10.1016/j.urolonc.2005.01.002. PMID 16144667
- [Background] Fowke JH, Signorello LB, Underwood W 3rd, Ukoli FA, Blot WJ. Obesity and prostate cancer screening among African-American and Caucasian men. Prostate. 2006 Sep 15;66(13):1371-80. doi: 10.1002/pros.20377. PMID 16752375
- [Background] Murff HJ, Peterson NB, Fowke JH, Hargreaves M, Signorello LB, Dittus RS, Zheng W, Blot WJ. Colonoscopy screening in African Americans and Whites with affected first-degree relatives. Arch Intern Med. 2008 Mar 24;168(6):625-31. doi: 10.1001/archinte.168.6.625. PMID 18362255
- [Background] Barocas DA, Gray DT, Fowke JH, Mercaldo ND, Blume JD, Chang SS, Cookson MS, Smith JA Jr, Penson DF. Racial variation in the quality of surgical care for prostate cancer. J Urol. 2012 Oct;188(4):1279-85. doi: 10.1016/j.juro.2012.06.037. Epub 2012 Aug 16. PMID 22902011
- [Background] Barocas DA, Grubb R 3rd, Black A, Penson DF, Fowke JH, Andriole G, Crawford ED. Association between race and follow-up diagnostic care after a positive prostate cancer screening test in the prostate, lung, colorectal, and ovarian cancer screening trial. Cancer. 2013 Jun 15;119(12):2223-9. doi: 10.1002/cncr.28042. Epub 2013 Apr 4. PMID 23559420
- [Background] Mandal DM, Sartor O, Halton SL, Mercante DE, Bailey-Wilson JE, Rayford W. Recruitment strategies and comparison of prostate cancer-specific clinical data on African-American and Caucasian males with and without family history. Prostate Cancer Prostatic Dis. 2008;11(3):274-9. doi: 10.1038/pcan.2008.5. Epub 2008 Feb 12. PMID 18268528
- [Background] Carpenter WR, Godley PA, Clark JA, Talcott JA, Finnegan T, Mishel M, Bensen J, Rayford W, Su LJ, Fontham ET, Mohler JL. Racial differences in trust and regular source of patient care and the implications for prostate cancer screening use. Cancer. 2009 Nov 1;115(21):5048-59. doi: 10.1002/cncr.24539. PMID 19637357
- [Background] Rayford W. Managing the low-socioeconomic-status prostate cancer patient. J Natl Med Assoc. 2006 Apr;98(4):521-30. PMID 16623064
- [Background] McHorney CA, Ware JE Jr, Lu JF, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. Med Care. 1994 Jan;32(1):40-66. doi: 10.1097/00005650-199401000-00004. PMID 8277801

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Navigation | Brochure
Started | 905 | 1746 | 1800
Completed | 905 | 1746 | 1800
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Reference group N=905
- Navigation: Phone calls done by Research Educator N=1746
- Brochure: Education through sending brochures to study participants N=1800
- Total: Total of all reporting groups
Arm/Group | Control | Navigation | Brochure | Total
Number analyzed (Participants) | 905 | 1746 | 1800 | 4451
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.94 (8.76) | 65.35 (8.62) | 65.78 (8.72) | 65.64 (8.69)
Age, Customized [Count of Participants; unit: Participants]
  50 to 65 years | 405 | 842 | 839 | 2086
  65 years plus | 500 | 907 | 958 | 2365
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 520 | 1028 | 1025 | 2573
  Male | 385 | 718 | 775 | 1878
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Americans | 905 | 1746 | 1800 | 4451

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Yield
Description: measured by the proportion of targeted survivors who, at the time of the recruitment call, after the screening process is complete, decide to participate in AMPLIFI.
Time Frame: within 3 months of receiving intervention
Population: Number of participants analyzed is equal to survivors eligible for the AMPLIFI trial
Measure: Number; unit: participants
Arm/Group | Control | Navigation | Brochure
Number analyzed (Participants) | 37 | 70 | 73
participants | 13 | 33 | 37
Statistical Analysis 1: Comparison: Control vs Navigation; Test type: Superiority; p = 0.2345, Regression, Logistic; Odds Ratio (OR) = 1.647, 95% CI 2-sided [0.724 to 3.746]
Statistical Analysis 2: Comparison: Control vs Brochure; Test type: Superiority; p = 0.124, Regression, Logistic; Odds Ratio (OR) = 1.897, 95% CI 2-sided [0.839 to 4.291]

2. Post Hoc Outcome: Survivors Reached by Recruiter
Description: Proportion of targeted survivors who were reached by phone by an AMPLIFI study recruiter
Time Frame: within 3 months of the AWEI intervention
Population: All randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Navigation | Brochure
Number analyzed (Participants) | 905 | 1746 | 1800
Participants | 363 | 659 | 688
Statistical Analysis 1: Comparison: Control Group vs Navigation; Test type: Superiority; p = 0.2352, Regression, Logistic; Odds Ratio (OR) = 0.905, 95% CI 2-sided [0.768 to 1.067]
Statistical Analysis 2: Comparison: Control Group vs Brochure; Test type: Superiority; p = 0.3418, Regression, Logistic; Odds Ratio (OR) = 0.924, 95% CI 2-sided [0.785 to 1.088]

3. Post Hoc Outcome: Screened
Description: Proportion of survivors reached by a recruiter who were screened for eligibility
Time Frame: within 3 months of the AWEI intervention
Population: Survivors reached by the recruiter
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Navigation | Brochure
Number analyzed (Participants) | 363 | 659 | 688
Participants | 100 | 208 | 218
Statistical Analysis 1: Comparison: Control Group vs Brochure; Test type: Superiority; p = 0.1653, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.921 to 1.615]
Statistical Analysis 2: Comparison: Control Group vs Navigation; Test type: Superiority; p = 0.181, Regression, Logistic; Odds Ratio (OR) = 1.213, 95% CI 2-sided [0.914 to 1.609]

ADVERSE EVENTS:
Time Frame: No adverse events were monitored
Description: Total Number of Participants at Risk (e.g., "All-Cause Mortality, Serious, and Other [Not Including Serious] is 0 because Adverse Events were not monitored/assessed due to the minimal risk interventions tested
Arm/Group | Control | Navigation | Brochure
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT04683510/Prot_SAP_000.pdf